CLINICAL TRIAL: NCT00101088
Title: A Phase I Study of CCI-779 in Combination With Imatinib Mesylate in Chronic Myelogenous Leukemia
Brief Title: Temsirolimus and Imatinib Mesylate in Treating Patients With Chronic Myelogenous Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00073; UCI-04-04; R21CA112936 (NIH)
Record Dates: First submitted 2005-01-07; First posted 2005-01-10 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Blastic Phase Chronic Myelogenous Leukemia; Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Chronic Phase Chronic Myelogenous Leukemia; Relapsing Chronic Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase | interventions — Imatinib Mesylate; temsirolimus; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (imatinib mesylate, temsirolimus) (Experimental): Patients receive temsirolimus IV over 30 minutes once on days 1, 8, 15, and 22 and oral imatinib mesylate once daily on days 1-28. Courses repeat every 28 days in the absence of unacceptable toxicity or disease progression
  Interventions: Drug: imatinib mesylate; Drug: temsirolimus; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: imatinib mesylate — Given orally
  Other Names: CGP 57148; Gleevec; Glivec
Drug: temsirolimus — Given IV
  Other Names: CCI-779; cell cycle inhibitor 779; Torisel
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of temsirolimus when given with imatinib mesylate in treating patients with chronic myelogenous leukemia. Drugs used in chemotherapy, such as temsirolimus, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Imatinib mesylate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving temsirolimus with imatinib mesylate may kill more cancer cells

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the safety and tolerability of temsirolimus when administered with imatinib mesylate in patients with chronic myelogenous leukemia.

II. Determine potential dose-limiting toxic effects of this regimen in these patients.

III. Determine, preliminarily, hematologic and cytogenetic response rates in patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of temsirolimus.

Patients receive temsirolimus intravenously (IV) over 30 minutes once on days 1, 8, 15, and 22 and oral imatinib mesylate once daily on days 1-28. Courses repeat every 28 days in the absence of unacceptable toxicity or disease progression. Patients receive 2 additional courses beyond maximal response. Cohorts of 3-6 patients receive escalating doses of temsirolimus until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed for survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed chronic myelogenous leukemia (CML)

  * Philadelphia chromosome-positive OR Bcr-Abl-positive disease, meeting 1 of the following criteria:

    * Accelerated phase, defined by at least 1 of the following:

      * 10-19% blasts in the peripheral blood or bone marrow
      * At least 20% basophils in peripheral blood or bone marrow
      * Platelet count < 100,000/mm^3 (unrelated to therapy)
      * Platelet count > 1,000,000/mm^3 (unresponsive to therapy)
      * Increasing splenomegaly AND increasing WBC count (unresponsive to therapy)
      * Clonal evolution
    * Blast phase, defined by 1 of the following:

      * At least 20% blasts in peripheral blood or bone marrow
      * Extramedullary disease
    * Chronic phase, defined by all of the following:

      * Less than 10% blasts in peripheral blood or bone marrow
      * Less than 20% basophils in peripheral blood or bone marrow
      * Platelet count > 100,000/mm^3
      * Absence of clonal evolution
* May have received and/or failed prior imatinib mesylate therapy

  * Patients not previously treated with imatinib mesylate receive oral imatinib mesylate once daily 14 days before beginning study drug

    * Must be able to tolerate 600 mg per day of imatinib mesylate before starting CCI-779
  * Patients with chronic phase disease must have failed prior imatinib mesylate at a dose ≥ 600 mg/day, as defined by 1 of the following:

    * Must not have achieved or must have lost hematologic response within 3 months after the start of imatinib mesylate
    * Must not have achieved or must have lost cytogenetic response after 6 months of treatment with imatinib mesylate
    * Must not have achieved or must have lost major cytogenetic response after 12 months of treatment with imatinib mesylate
    * Must have lost complete cytogenetic response
* Bone marrow aspirate and biopsy with cytogenetics and fluorescent in situ hybridization confirming t(9;22) completed within the past 28 days
* Performance status - SWOG 0-2
* More than 3 months
* See Disease Characteristics
* Bilirubin normal
* AST and ALT < 2.5 times upper limit of normal (ULN) (5 times ULN if suspected liver involvement with leukemia)
* Creatinine normal
* Creatinine clearance > 60 mL/min
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Ejection fraction ≥ 50% by echocardiogram or MUGA scan for patients with known positive cardiac history (e.g., heart failure, coronary artery disease, cardiomegaly on prior chest x-ray, or valvular heart disease)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Fasting cholesterol ≤ 350 mg/dL
* Fasting triglycerides ≤ 400 mg/dL
* No history of allergic reaction attributed to compounds of similar chemical or biologic composition to temsirolimus or imatinib mesylate
* No active or ongoing infection
* No psychiatric illness or social situation that would preclude study compliance
* No other active malignancy except nonmelanoma skin cancer
* No other uncontrolled illness
* At least 48 hours since prior interferon alfa for CML
* At least 6 weeks since prior stem cell transplantation
* No concurrent biologic agents
* No concurrent prophylactic colony-stimulating factors
* At least 24 hours since prior hydroxyurea for CML
* At least 7 days since prior mercaptopurine or vinca alkaloids for CML
* At least 7 days since prior low-dose cytarabine (< 30 mg/m^2 every 12-24 hours) for CML
* At least 14 days since prior homoharringtonine for CML
* At least 14 days since prior moderate-dose cytarabine (100-200 mg/m^2 for 5-7 days) for CML
* At least 21 days since prior anthracyclines, mitoxantrone, cyclophosphamide, etoposide, or methotrexate for CML
* At least 28 days since prior high-dose cytarabine (1-3 g/m^2 every 12-24 hours for 6-12 doses) for CML
* At least 6 weeks since prior busulfan for CML
* No concurrent hydroxyurea
* No other concurrent chemotherapy
* At least 7 days since prior steroids for CML
* No prior organ transplantation
* More than 2 weeks since prior major surgery (e.g., thoracotomy or intra-abdominal surgery)
* Recovered from all prior therapy
* Prior experimental therapy allowed provided completion of treatment corresponds to a duration > 5 half-lives of the experimental drug or any known active metabolite before study
* No concurrent cyclosporine
* No concurrent anagrelide
* No concurrent oral anticoagulants, including warfarin
* No concurrent CYP3A4 inducers or inhibitors
* No concurrent tacrolimus
* No concurrent plasmapheresis
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No other concurrent anticancer therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2005-04; Primary Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Unacceptable toxicity graded according to the NCI CTCAE version 3.0 | Up to 5 years

SECONDARY OUTCOMES:
Disease progression | Up to 5 years
Duration of response | Up to 5 years
  Presented using descriptive statistics.
Survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Tiong Ong, Principal Investigator — University of California Medical Center At Irvine-Orange Campus
Locations (1):
- University of California Medical Center At Irvine-Orange Campus, Orange, California, United States